CLINICAL TRIAL: NCT00488618
Title: A Double-Blind, Placebo-Controlled Evaluation of the Safety and Efficacy of RGH-188 in Patients With Acute Mania Associated With Bipolar I Disorder
Brief Title: Study Evaluating Cariprazine (RGH-188) in the Treatment of Patients With Acute Mania
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Collaborators: Gedeon Richter Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RGH-MD-31
Record Dates: First submitted 2007-06-19; First posted 2007-06-20 (Estimated); Results first posted 2017-04-14 (Actual); Last update posted 2017-04-14 (Actual); Status verified 2017-03

CONDITIONS: Bipolar Disorder
Keywords: Mania; Bipolar I Disorder; Acute Mania Associated with Bipolar I Disorder
MeSH Terms: conditions — Bipolar Disorder; Mania | interventions — cariprazine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cariprazine (Experimental): Cariprazine 3 mg - 12 mg capsules oral administration, once per day for 3 weeks.
  Interventions: Drug: Cariprazine (RGH-188)
- Placebo (Placebo Comparator): Placebo dose-matching cariprazine capsules oral administration, once per day for 3 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cariprazine (RGH-188) — Cariprazine 3 mg - 12 mg oral administration, once per day.
  Arms: Cariprazine
Drug: Placebo — Dose-matched placebo oral administration, once per day.
  Arms: Placebo

SUMMARY:
This is a study designed to evaluate the efficacy, safety, and tolerability of RGH-188 monotherapy in the treatment of acute mania. This study will be 5 weeks in duration; 3 weeks double-blind treatment and 2-weeks safety follow-up. All patients meeting the eligibility criteria will be randomized to one of two treatment groups: RGH-188 or placebo

ELIGIBILITY:
Inclusion Criteria:

* Male or female inpatients 18 to 65 years of age
* Meeting Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV) criteria for bipolar I disorder, acute manic or mixed episode
* Having a total Young Mania Rating Scale (YMRS) score >= 20 and a score of at least 4 on two of the following YMRS items:

  * Irritability,
  * Speech,
  * Content, and
  * Disruptive/Aggressive Behavior

Exclusion Criteria:

* Patients who exhibit abnormalities on physical examination, have abnormal vital-signs, electrocardiogram (ECG), or clinical laboratory values [such as thyroid-stimulating hormone (TSH)].
* Patients with Montgomery-Åsberg Depression Rating Scale (MADRS) total score >= 18 at Visit 2.
* Patients experiencing first manic episode.
* Patients that have received electroconvulsive therapy (ECT) or a depot neuroleptic in the 3 months prior to Visit 1.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2007-06; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- For information regarding investigative sites, contact Forest Professional Affairs, St Louis, Missouri, United States

REFERENCES:
- [Derived] McIntyre RS, Masand PS, Earley W, Patel M. Cariprazine for the treatment of bipolar mania with mixed features: A post hoc pooled analysis of 3 trials. J Affect Disord. 2019 Oct 1;257:600-606. doi: 10.1016/j.jad.2019.07.020. Epub 2019 Jul 5. PMID 31344528
- [Derived] Earley W, Durgam S, Lu K, Ruth A, Nemeth G, Laszlovszky I, Yatham LN. Clinically relevant response and remission outcomes in cariprazine-treated patients with bipolar I disorder. J Affect Disord. 2018 Jan 15;226:239-244. doi: 10.1016/j.jad.2017.09.040. Epub 2017 Sep 25. PMID 29017067

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Cariprazine
Started | 120 | 118
Safety Population: Received Study Drug | 118 | 118
Completed | 73 | 75
Not Completed | 47 | 43
Not completed — Adverse Event | 13 | 17
Not completed — Insufficient Therapeutic Response | 18 | 11
Not completed — Protocol Violation | 0 | 2
Not completed — Withdrawal of Consent | 15 | 13
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Cariprazine | Total
Number analyzed (Participants) | 118 | 118 | 236
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.7 (11.0) | 38.0 (10.3) | 38.3 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 38 | 79
  Male | 77 | 80 | 157
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 10
  Not Hispanic or Latino | 114 | 112 | 226
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 55 | 47 | 102
  Black | 31 | 36 | 67
  Asian | 28 | 30 | 58
  Other | 4 | 5 | 9
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 79.3 (20.0) | 75.0 (20.3) | 77.2 (20.2)
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 170.0 (10.4) | 169.9 (10.0) | 170.0 (10.2)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/meter(m)^2] | 27.2 (5.8) | 25.8 (5.9) | 26.5 (5.9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Young Mania Rating Scale (YMRS) Total Score at Week 3
Description: The YMRS is an 11-item scale that assesses manic symptoms based on the participant's perception of his or her condition over the previous 48 hours, as well as the physician's clinical observations during the interview. The 11-items are elevated mood, increased motor activity-energy, sexual interest, sleep, irritability, rate and amount of speech, language-thought disorder, content, disruptive-aggressive behavior, appearance, and insight. The severity of the abnormality for 7-items are rated on a five-point scale (0-4) and 4-items on a nine-point scale (0-8). The individual scores are summed for a total possible score of 0 (best) to 60 (worst). A negative change from Baseline indicates improvement. Analyses are based on an Analysis of Covariance (ANCOVA) model for change from Baseline with treatment group and study center as factors and Baseline value as covariate.
Time Frame: Baseline, Week 3
Population: Intent-to-treat Population included Participants who received at least 1 dose of study drug and who had at least 1 post-baseline YMRS assessment, last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Cariprazine
Number analyzed (Participants) | 117 | 118
score on a scale | -8.91 (1.083) | -15.02 (1.078)
Statistical Analysis 1: Comparison: Placebo vs Cariprazine; Test type: Superiority or Other; p < 0.0001, ANCOVA; Least Squares Mean Difference = -6.1, 95% CI 2-sided [-8.9 to -3.3] — cariprazine - placebo

2. Secondary Outcome: Change From Baseline in Clinical Global Impression-Severity (CGI-S) Total Score at Week 3
Description: The CGI-S measures the investigator's assessment of overall severity of the participant's illness compared with the severity of illness in other patients the physician has observed using a 7-point scale (1=Normal, not ill at all to 7=Among the most extremely ill participants). A negative change from Baseline indicates improvement. Analyses are based on ANCOVA model for change from Baseline with treatment group and study center as factors and Baseline CGI-S score as covariate.
Time Frame: Baseline, 3 Weeks
Population: Intent-to-treat Population included all participants who received at least 1 dose of study drug and who had at least 1 post-baseline YMRS assessment, LOCF.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Cariprazine
Number analyzed (Participants) | 117 | 118
score on a scale | -0.93 (0.125) | -1.57 (0.125)
Statistical Analysis 1: Comparison: Placebo vs Cariprazine; Test type: Superiority or Other; p = 0.0001, ANCOVA; Least Squares Mean Difference = -0.64, 95% CI 2-sided [-0.97 to -0.32] — cariprazine - placebo

ADVERSE EVENTS:
Time Frame: First dose of study drug to 30 days past last dose (Up to 51 days)
Description: Safety Population included all participants who received at least 1 dose of study drug.
Arm/Group | Placebo | Cariprazine
Serious Adverse Events (participants affected / at risk) | 6/118 | 7/118
Other Adverse Events (participants affected / at risk) | 73/118 | 90/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=118) | Cariprazine (N=118)
Mania (Psychiatric disorders) | 5 | 4
Convulsion (Nervous system disorders) | 0 | 1
Extrapyramidal disorder (Nervous system disorders) | 0 | 1
Delusion (Psychiatric disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=118) | Cariprazine (N=118)
Vision blurred (Eye disorders) | 1 | 7
Constipation (Gastrointestinal disorders) | 10 | 19
Nausea (Gastrointestinal disorders) | 12 | 19
Dyspepsia (Gastrointestinal disorders) | 9 | 15
Vomiting (Gastrointestinal disorders) | 6 | 10
Diarrhoea (Gastrointestinal disorders) | 9 | 8
Toothache (Gastrointestinal disorders) | 8 | 3
Pyrexia (General disorders) | 7 | 8
Blood creatine phosphokinase increased (Investigations) | 6 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 6
Extrapyramidal disorder (Nervous system disorders) | 13 | 29
Headache (Nervous system disorders) | 26 | 24
Akathisia (Nervous system disorders) | 8 | 23
Dizziness (Nervous system disorders) | 8 | 12
Sedation (Nervous system disorders) | 2 | 7
Tremor (Nervous system disorders) | 6 | 6
Insomnia (Psychiatric disorders) | 3 | 10
Restlessness (Psychiatric disorders) | 1 | 8
Agitation (Psychiatric disorders) | 10 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study will be the property of Forest Research Institute, Inc. An integrated clinical and statistical report will be prepared at the completion of the study.

Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and Forest Research Institute, Inc.